CLINICAL TRIAL: NCT04864561
Title: A Randomized, Observer-Blind, Controlled, Superiority Study To Compare The Immunogenicity Against COVID-19, Of VLA2001 Vaccine To AZD1222 Vaccine, In Adults Including a Randomized, Observer-blind, Placebo Controlled Part in Adolescents (≥12 to <18 Years)
Brief Title: COV-COMPARE Immunogenicity of Vaccine VLA2001 Compared to AZD1222
Acronym: COV-COMPARE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Valneva Austria GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: VLA2001-301
Record Dates: First submitted 2021-04-23; First posted 2021-04-29 (Actual); Last update posted 2023-03-20 (Actual); Status verified 2023-03

CONDITIONS: SARS-CoV-2 Virus Infection
Keywords: VLA2001; SARS-CoV-2 Virus Infection; COVID-19; inactivated-adjuvanted SARS-CoV-2 virus vaccine
MeSH Terms: conditions — COVID-19 | interventions — VLA2001 COVID-19 vaccine; ChAdOx1 nCoV-19

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: study participants aged 18-29 years at the time of enrolment are unblinded, study participant aged 12-18 and 30 years above at the time of enrolment are blinded (sentinel group is unblinded) until 28 days after vaccination on day 208, when all participants will be unblinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- VLA2001 (Experimental): <30 years will receive VLA2001; participants aged ≥30 years will be randomised 2:1 to receive VLA2001 or AZD1222
  Interventions: Biological: VLA2001
- AZD1222 (Active Comparator): <30 years will receive VLA2001; participants aged ≥30 years will be randomised 2:1 to receive VLA2001 or AZD1222
  Interventions: Biological: AZD1222
- VLA2001 - adolescent part (Experimental): ≥12 to < 18 years will be randomized 1:1 to receive VLA2001 or Placebo
  Interventions: Biological: VLA2001 - adolescent part
- Placebo (Placebo Comparator): ≥12 to < 18 years will be randomized 1:1 to receive VLA2001 or Placebo
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: VLA2001 — whole virus inactivated SARS-CoV-2 vaccine adjuvanted with cytosine phospho-guanine (CpG) 1018 in combination with aluminium hydroxide 2 vaccinations 28 days apart
  Arms: VLA2001
Biological: AZD1222 — 2 vaccinations 28 days apart AZD1222 is a recombinant, replication-defective chimpanzee adenovirus expressing the SARS-CoV-2 S surface glycoprotein.
  Arms: AZD1222
Biological: VLA2001 - adolescent part — whole virus inactivated SARS-CoV-2 vaccine adjuvanted with cytosine phospho-guanine (CpG) 1018 in combination with aluminium hydroxid 2 vaccinations 28 days apart and with a booster vaccination on day 208. Placebo group will receive VLA2001 on day 208 and following second vaccination 28 days later.
  Arms: VLA2001 - adolescent part
Biological: Placebo — 2 vaccinations 28 days apart with placebo (PBS buffer based on Dulbecco's PBS media formulation without Calcium and Magnesium )
  Arms: Placebo

SUMMARY:
This is a multicentre, randomized, observer-blind, active-controlled, superiority, study in adults to compare the immunogenicity of VLA2001 to AZD1222 in terms of GMT of SARS-CoV-2-specific neutralising antibodies. Furthermore, VLA2001 will be compared to placebo in an adolescent population.

DETAILED DESCRIPTION:
Approximately 4000 Adult participants will be recruited in the study. About 3000 participants aged 30 years and above will be randomized in a 2:1 ratio to receive 2 intramuscular recommended doses of either VLA2001 (n=2000) or AZD1222 (n=1000). In addition, approximately 1000 subjects aged 18-29 years will participate in this study in a non-randomized, open-label fashion to receive VLA2001. The 2 doses of vaccination for both vaccines will be administered 28 days apart, on Days 1 and 29. All visits will be conducted at the clinical site on an outpatient basis.

All participants - except those who already received a licensed COVID-19 vaccine outside of the study - will be offered a booster dose with VLA2001 between Jan and Mar 2022 and will have a follow-up visit 14 days (Visit B2) and 6months after the booster dose.

Approximately 660 Adolescent participants were planned to be recruited and randomized in a 1:1 ratio to receive 2 intramuscular doses of either VLA2001 (n=330) or placebo (n=300). Participants in the placebo group will receive a 2-dose primary immunization with VLA2001 on Day 85 and the second vaccination 28 days later. For safety reasons, the first 16 adolescents will be enrolled in an open label, non-randomized manner (sentinel dosing).

Recruitment of adolescent participants has been stopped after recruitment of 6 randomized participants (3 randomized to VLA2001 and 3 participants randomized to placebo) due to the low recruitment rate. The study design ensures a safety follow-up of at least 6 months after the last VLA2001 vaccination/booster for all enrolled study participants

Participants will be provided with an electronic Diary (e-Diary) and will be trained to record specifically solicited systemic and local symptoms daily as well as any additional AEs during follow-up period after each of both vaccinations up to the next visit to the site until Day 43 visit has been completed.

ELIGIBILITY:
Inclusion Criteria:

1. Participants must have read, understood, and signed the informed consent form (ICF).
2. Participants of either gender aged 12 years and older at screening.
3. Medically stable
4. Must be able to attend all visits of the study and comply with all study procedures,
5. Women of childbearing potential (WOCBP) must be able and willing to use at least 1 highly effective method of contraception for a minimum of 3 months after the last dose of study vaccine.
6. WOCBPs must have a negative pregnancy test prior to each vaccination.

Exclusion Criteria:

1. Participant is pregnant or planning to become pregnant within 3 months after study vaccine administration.
2. History of allergy to any component of the vaccine.
3. Significant infection (e.g. positive SARS-CoV-2 RT-PCR) or other acute illness, including fever > 100 °F (> 37.8 °C) 48 hours before vaccination.
4. Participant has a known or suspected defect of the immune system
5. Participant has a history of cerebral venous sinus thrombosis, heparin-induced thrombocytopenia or antiphospholipid syndrome.
6. Participant has a history of malignancy in the past 5 years other than squamous cell or basal cell skin cancer. If there has been surgical excision or treatment more than 5 years ago that is considered to have achieved a cure, the participant may be enrolled. A history of hematologic malignancy is a permanent exclusion. Participants with a history of skin cancer must not be vaccinated at the previous tumour site.
7. History of drug dependency or current use of drug of abuse or alcohol abuse at screening.
8. Significant blood loss (> 450 mL) or has donated 1 or more units of blood or plasma within 6 weeks prior to the expected day of randomization (Visit 1).
9. History of clinically significant bleeding disorder, or prior history of significant bleeding or bruising following IM injections or venepuncture.
10. Severe and uncontrolled ongoing autoimmune or inflammatory disease History of Guillain-Barre syndrome or any other demyelinating condition.
11. Any other significant disease, disorder or finding which in the opinion of the investigator may significantly increase the risk to the volunteer

    Prior/concomitant therapy:
12. Receipt of immunoglobulin or another blood product within the 3 months before expected day of randomization (visit 1) in this study or those who expect to receive immunoglobulin or another blood product during this study.
13. Receipt of medications and or vaccinations intended to prevent COVID-19.
14. Receipt of any vaccine (licensed or investigational), other than licensed influenza vaccine, within 28 days prior to the expected day of randomization (Visit 1).
15. Any member of the study team or sponsor.
16. An immediate family member or household member of the study's personnel.

Booster Vaccination (Adults and Adolescents)

In addition to the above-described eligibility criteria, the following criteria must be met:

1. Participant has not received another licensed COVID-19 vaccine during the study

Min Age: 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 4034 (Actual)
Dates: Start 2021-04-26 (Actual); Primary Completion 2021-07-19 (Actual); Study Completion 2023-03-13 (Actual)

PRIMARY OUTCOMES:
Immune response measured after completion of a 2-dose immunization schedule, as determined by the geometric mean titer (GMT) ratio in adults and GMT in adolescents of SARS-CoV-2-specific neutralizing antibodies | Day 43
Immune response measured after completion of a 2-dose immunization schedule, as determined by Seroconversion in adults and adolescents (definded as 4-fold increase from baseline) of SARS-CoV-2-specific neutralizing antibodies | Day 43
Frequency and severity of any Adverse Events (AE) | Up to Day 43 post-vaccination

SECONDARY OUTCOMES:
Proportion of adult participants with seroconversion | on Day 8 (age 55+ only), Day 29, Day 71 and Day 208
  Seroconversion is defined as >= 4-fold increase in SARS-CoV-2 neutralizing antibody titer against the Wuhan strain and IgG antibodies directed against the S-protein of the Wuhan strain between Day 1 and the defined post-vaccination timepoints
Proportion of adolescent participants with Seroconversion | on Day 43, Day 71/Day 85 and Day 127
Immune response in adults as determined geometric mean titer (GMT) of SARS-CoV-2-specific neutralising antibodies | on Day 8 (age 55+ only), Day 29, Day 71 and Day 208
Immune response in adolescents as determined by the GMT of SARS-CoV-2-specific neutralising antibodies | on Day 43, Day 71/Day 85 and Day 127
GMT ratio of SARS-CoV-2-specific neutralizing antibodies in the adolescent and adult population | on Day 43
Immune response in adults determined by the GMT of IgG antibodies to SARS-CoV-2 S-protein | on Day 8 (age 55+ only), Day 29, Day 43, Day 71 and Day 208
Immune response in adolescents determined by the GMT of IgG antibodies to SARS-CoV-2 S-protein | on Day 43, Day 71/Day 85 and Day 127
GMT ratio of IgG antibodies to SARS-CoV-2 S-protein in the adolescent and adult population | on Day 43
Assessment of T-cell responses from PBMCs on selected time points in a subset of participants after in vitro stimulation with SARS-CoV-2 antigens using e.g., ELISpot or intracellular cytokine staining | Adult: Day 29, Day 43, Day 71 and Day 208, Adolescence: on Day 43, Day 71/Day 85 and Day 127
Frequency and severity of solicited injection site and systemic reactions | until 7 days after each and any vaccination
Frequency and severity of any AE | through study completion, up to 13 or 16 months
Frequency and severity of any unsolicited AE | through study completion, up to 13 or 16 months
Frequency and severity of any unsolicited vaccine-related AE | through study completion, up to 13 or 16 months
Frequency and severity of any serious adverse event (SAE) | through study completion, up to 13 or 16 months
Frequency and severity of any adverse event of special interest (AESI) | through study completion, up to 13 or 16 months
Geometric mean fold rise (GMFR) with regards to SARS-CoV-2-specific neutralizing antibodies | from day of booster vaccination to 14 days after booster vaccination
  adult participants with single booster
GMT of SARS-CoV-2-specific neutralizing antibodies as measured by MNA50 including formal non-inferiority testing on the GMT ratio | on day of booster vaccination, 14 days and 6 months post booster
  adult participants with single booster
Proportion of participants with 4-fold increase with regards to SARS-CoV-2-specific neutralizing antibodies | from day of booster vaccination to 14 days after booster vaccination
  adult participants with single booster
GMFR with regards to S-protein binding antibodies | from day of booster vaccination to 14 days after booster vaccination
  adult participants with single booster
Proportion of participants with 4-fold increase with regards to S-protein binding antibodies | from day of booster vaccination to 14 days after booster vaccination
  adult participants with single booster
Assessment of T-cell responses from PBMCs in a subset of participants after in vitro stimulation with SARS-CoV-2 antigens using ELISpot | on day of booster vaccination, 14 days and 6 months post booster
  adult participants with single booster
Frequency and severity of solicited injection site and systemic reactions | 7 days after booster vaccination
  adult participants with single booster
Frequency and severity of any unsolicited AE | up to 6 months after booster dose
  adult participants with single booster
Frequency and severity of any vaccine-related | up to 6 months after booster dose
  adult participants with single booster
Frequency and severity of any serious adverse event (SAE) | up to 6 months after booster dose
  adult participants with single booster
Frequency and severity of any adverse event of special interest (AESI) | up to 6 months after booster dose
  adult participants with single booster
Geometric mean fold rise (GMFR) with regards to SARS-CoV-2-specific neutralizing antibodies | from day of booster vaccination to 14 days after booster vaccination
  adolescent participants with single booster
GMT of SARS-CoV-2-specific neutralizing antibodies as measured by MNA50 | Day of booser vaccination and 14 days post booster
  adolescent participants with single booster
Proportion of participants with 4-fold increase with regards to SARS-CoV-2-specific neutralizing antibodies | from day of booster vaccination to 14 days after booster vaccination
  adolescent participants with single booster
GMFR with regards to S-protein binding antibodies | from day of booster vaccination to 14 days after booster vaccination
  adolescent participants with single booster
Proportion of participants with 4-fold increase with regards to S-protein binding antibodies | from day of booster vaccination to 14 days after booster vaccination
  adolescent participants with single booster
GMT measured as IgG antibodies against SARS-CoV-2 as determined by ELISA | Day of booser vaccination and 14 days post booster
  adolescent participants with single booster
Assessment of T-cell responses from PBMCs in a subset of participants after in vitro stimulation with SARS-CoV-2 antigens using ELISpot | Day of booser vaccination and 14 days post booster
  adolescent participants with single booster
Frequency and severity of solicited injection site and systemic reactions | up to 7 days after booster vaccination
  adolescent participants with single booster
Frequency and severity of any unsolicited AE | 180 days post booster vaccination
  adolescent participants with single booster
Frequency and severity of any serious adverse event (SAE) | 180 days post booster vaccination
  adolescent participants with single booster
Frequency and severity of any adverse event of special interest (AESI) | 180 days post booster vaccination
  adolescent participants with single booster
GMT measured as IgG antibodies against SARS-CoV-2 as determined by ELISA | on day of booster vaccination, 14 days and 6 months post booster
  adult participants with single booster
Frequency and severity of any vaccine related AE | 180 days post booster vaccination
  adolescent participants with single booster

CONTACTS AND LOCATIONS:
Overall Officials: Valneva Clinical Development, Study Chair — Valneva Austria GmbH
Locations (31):
- United Kingdom (31):
  - Barnsley Hospital NHS FT, Barnsley
  - University Hospitals Birmingham NHS Foundation Trust, Birmingham
  - Blackpool Teaching Hospitals NHS Foundation Trust, Blackpool
  - North Bristol NHS Trust, Bristol
  - University Hospitals Bristol and Weston NHS Foundation Trust, Bristol
  - Cambridge Biomedical Research Centre, Cambridge
  - Cheadle Community Hospital, Cheadle
  - University Hospitals Coventry & Warwickshire, Coventry
  - Western General Hospital, Edinburgh - NHS Lothian, Edinburgh
  - Epsom and St. Helier University Hospitals NHS Trust, Epsom
  - Queen Elizabeth University Hospital-Glasgow- NHS Greater Glasgow, Glasgow
  - Royal Surrey County Hospital NHS Foundation Trust, Guildford
  - University Hospitals of Leicester NHS Trust, Leicester
  - NHS Foundation Trust Royal Liverpool University Hospital, Liverpool
  - Barts Health NHS Trust, London
  - Panthera London, London
  - Royal Free London NHS Foundation Trust, London
  - King's College Hospital, Trust College HOspital NHS Foundation Trust, London
  - Chelsea and Westminster Hospital NHS Trust, London
  - St George's University Hospitals NHS Foundation Trust, London
  - NIHR UCLH Clinical Research Facility, London
  - The Newcastle upon Tyne Hospitals NHS Foundation Trust, Freeman Hospital Newcastle, Newcastle
  - Northumbria Healthcare NHS Foundation Trust - North Tyneside General Hospital, North Shields
  - Lakeside Healthcare Research, Northampton
  - Nottingham University Hospitals NHS Trust, Nottingham
  - University Hospital Plymouth NHS Trust, Plymouth
  - Panthera Biopartners Preston, Preston
  - Panthera Biopartners Manchester, Rochdale
  - Northern Care Alliance NHS Group, Salford Royal NHS Foundation Trust, Salford
  - Southampton University Hospitals NHS Trust, Southampton
  - Royal Cornwall Hospitals NHS Trust, Truro

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Taucher C, Lazarus R, Dellago H, Maurer G, Weisova P, Corbic-Ramljak I, Dubischar K, Lilja A, Eder-Lingelbach S, Hochreiter R, Jaramillo JC, Junker H, Krammer M, Pusic P, Querton B, Larcher-Senn J, Hoffmann M, Pohlmann S, Finn A; Valneva Phase 3 Booster Trial Group. Safety and immunogenicity against ancestral, Delta and Omicron virus variants following a booster dose of an inactivated whole-virus COVID-19 vaccine (VLA2001): Interim analysis of an open-label extension of the randomized, controlled, phase 3 COV-COMPARE trial. J Infect. 2023 Sep;87(3):242-254. doi: 10.1016/j.jinf.2023.06.022. Epub 2023 Jul 3. PMID 37406777
- [Derived] Lazarus R, Querton B, Corbic Ramljak I, Dewasthaly S, Jaramillo JC, Dubischar K, Krammer M, Weisova P, Hochreiter R, Eder-Lingelbach S, Taucher C, Finn A; Valneva phase 3 trial group. Immunogenicity and safety of an inactivated whole-virus COVID-19 vaccine (VLA2001) compared with the adenoviral vector vaccine ChAdOx1-S in adults in the UK (COV-COMPARE): interim analysis of a randomised, controlled, phase 3, immunobridging trial. Lancet Infect Dis. 2022 Dec;22(12):1716-1727. doi: 10.1016/S1473-3099(22)00502-3. Epub 2022 Sep 5. PMID 36075233